CLINICAL TRIAL: NCT02091141
Title: My Pathway: An Open-Label Phase IIa Study Evaluating Trastuzumab/Pertuzumab, Erlotinib, Vemurafenib/Cobimetinib, Vismodegib, Alectinib, and Atezolizumab in Patients Who Have Advanced Solid Tumors With Mutations or Gene Expression Abnormalities Predictive of Response to One of These Agents
Brief Title: My Pathway: A Study Evaluating Herceptin/Perjeta, Tarceva, Zelboraf/Cotellic, Erivedge, Alecensa, and Tecentriq Treatment Targeted Against Certain Molecular Alterations in Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML28897; PRO 02 (Other: Genentech, Inc.)
Record Dates: First submitted 2014-03-17; First posted 2014-03-19 (Estimated); Results first posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-06

CONDITIONS: Neoplasms; Solid Tumors; Biliary Cancer; Salivary Cancer; Bladder Cancer
MeSH Terms: conditions — Neoplasms; Biliary Tract Neoplasms; Urinary Bladder Neoplasms | interventions — Trastuzumab; pertuzumab; Erlotinib Hydrochloride; Vemurafenib; cobimetinib; HhAntag691; alectinib; atezolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Trastuzumab Plus Pertuzumab (Experimental): Participants will receive trastuzumab 8 milligrams per kilogram (mg/kg) intravenous (IV) infusion as loading dose, followed by 6 mg/kg IV infusion every 3 weeks; and pertuzumab 840 mg IV infusion as loading dose, followed by 420 mg IV infusion every 3 weeks.
  Interventions: Drug: Trastuzumab; Drug: Pertuzumab
- Atezolizumab (Experimental): Participants will receive atezolizumab 1200 mg IV infusion every 3 weeks.
  Interventions: Drug: Atezolizumab
- Vemurafenib (Experimental): Participants will receive vemurafenib 960 mg orally twice daily (BID) in each 28-day cycle.
  Interventions: Drug: Vemurafenib
- Vemurafenib Plus Cobimetinib (Experimental): Participants will receive vemurafenib 960 mg orally twice daily (BID) in each 28-day cycle; and cobimetinib 60 mg orally once daily for 21 days on and 7 days off in each 28-day cycle.
  Interventions: Drug: Vemurafenib; Drug: Cobimetinib
- Vismodegib (Experimental): Participants will receive vismodegib 150 mg orally once daily in each 28-day cycle.
  Interventions: Drug: Vismodegib
- Alectinib (Experimental): Participants will receive alectinib 600 mg orally BID in each 28-day cycle.
  Interventions: Drug: Alectinib
- Erlotinib (Experimental): Participants will receive erlotinib 150 mg orally once daily in each 28-day cycle.
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Trastuzumab — Trastuzumab will be administered as per the schedule specified in the respective arm, until tumor progression or occurrence of unacceptable toxicity.
  Other Names: Herceptin
  Arms: Trastuzumab Plus Pertuzumab
Drug: Pertuzumab — Pertuzumab will be administered as per the schedule specified in the respective arm, until tumor progression or occurrence of unacceptable toxicity.
  Other Names: Perjeta
  Arms: Trastuzumab Plus Pertuzumab
Drug: Erlotinib — Erlotinib will be administered as per the schedule specified in the respective arm, until tumor progression or occurrence of unacceptable toxicity.
  Other Names: Tarceva
  Arms: Erlotinib
Drug: Vemurafenib — Vemurafenib will be administered as per the schedule specified in the respective arm, until tumor progression or occurrence of unacceptable toxicity.
  Other Names: Zelboraf
  Arms: Vemurafenib; Vemurafenib Plus Cobimetinib
Drug: Cobimetinib — Cobimetinib will be administered as per the schedule specified in the respective arm, until tumor progression or occurrence of unacceptable toxicity.
  Other Names: Cotellic
  Arms: Vemurafenib Plus Cobimetinib
Drug: Vismodegib — Vismodegib will be administered as per the schedule specified in the respective arm, until tumor progression or occurrence of unacceptable toxicity.
  Other Names: Erivedge
  Arms: Vismodegib
Drug: Alectinib — Alectinib will be administered as per the schedule specified in the respective arm, until tumor progression or occurrence of unacceptable toxicity.
  Other Names: Alecensa
  Arms: Alectinib
Drug: Atezolizumab — Atezolizumab will be administered as per the schedule specified in the respective arm, until tumor progression or occurrence of unacceptable toxicity.
  Other Names: Tecentriq
  Arms: Atezolizumab

SUMMARY:
This multicenter, non-randomized, open-label study will evaluate the efficacy and safety of six treatment regimens in participants with advanced solid tumors for whom therapies that will convey clinical benefit are not available and/or are not suitable options per the treating physician's judgment.

ELIGIBILITY:
General Inclusion Criteria:

* Life expectancy greater than or equal to (≥) 12 weeks
* Histologically documented metastatic cancer (solid tumors, not including hematologic malignancies)
* Participants who have received standard first-line therapy for metastatic cancer (except for the tumors for which no first-line therapy exists) and in whom a trial of targeted therapy is considered the best available treatment option. Eligible participants should not have available therapies that will convey clinical benefit and/or are not suitable options per the treating physician's judgment
* No previous treatment with the specific assigned study drug or any other drug sharing the same target
* Measurable disease by RECIST v1.1
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0 or 1 (For patients enrolling in the atezolizumab arm, ECOG score must be documented within 7 days prior to first treatment and confirmation of ECOG PS must be entered into the interactive web response system [IWRS] prior to initiation of treatment)
* Adequate hematologic, renal, and liver function as defined by the protocol
* If applicable, use of contraception methods or abstinence as defined by the protocol

Study-Drug Specific Inclusion Criteria:

Trastuzumab plus Pertuzumab

* Molecular testing results from clinical laboratory improvement amendments (CLIA)-certified laboratories (using tissue and/or blood) demonstrating HER2 overexpression or amplification. Participants must have one of the following tumor types: biliary cancer, salivary cancer, or bladder cancer

  a) For participants screened using a blood assay: obtain tissue-based testing result confirming study eligibility (within first 4 weeks after enrollment)
* Left ventricular ejection fraction (LVEF) greater than (>) 50 percent (%) or above the lower limit of the institutional normal range, whichever is lower
* Availability of an archival or new pre-treatment tissue sample is required if molecular testing was not performed by Foundation Medicine. Any available tumor tissue sample can be submitted. The tissue sample must be submitted within 4 weeks after enrollment

Erlotinib

* Molecular testing results from CLIA-certified laboratories (using tissue and/or blood) demonstrating epidermal growth factor receptor (EGFR)-activating mutations

Vemurafenib plus Cobimetinib

* Molecular testing results from CLIA-certified laboratories (using tissue and/or blood) demonstrating BRAF V600 mutations a) For participants screened using a blood assay: obtain tissue-based testing result confirming study eligibility (within first 4 weeks after enrollment)

Vismodegib

* Molecular testing results from CLIA-certified laboratories (using tissue and/or blood) demonstrating hedgehog pathway relevant mutation (activating mutation of smoothened [SMO] or loss-of-function mutation of protein patched homolog-1 [PTCH-1])

  a) For participants screened using a blood assay: obtain tissue-based testing result confirming study eligibility (within first 4 weeks after enrollment)
* All non-hematological adverse events related to any prior chemotherapy, surgery, or radiotherapy must have resolved to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Grade less than or equal to (≤) 2 prior to starting therapy

Alectinib

* Molecular testing results from CLIA-certified laboratories (using tissue and/or blood) demonstrating anaplastic lymphoma kinase (ALK) gene rearrangements, ALK mutations, ALK copy number gain or (for melanoma only) increased ALK expression or presence of ALK-alternative transcription initiation transcript (ALKATI) a) For participants screened using a blood assay: obtain tissue-based testing result confirming study eligibility (within first 4 weeks after enrollment)

Atezolizumab

* Molecular testing results from CLIA-certified laboratories (using tissue) demonstrating elevated tissue tumor mutational burden (tTMB ≥10 mutations/ Megabase [Mb])
* For patients where molecular testing was not performed using Foundation Medicine, submission of an archival or new pretreatment tissue sample is mandatory. For patients where molecular testing was performed using Foundation Medicine, submission of an archival or new pretreatment tissue sample is required, if available. The tissue sample must be submitted within 4 weeks after enrollment

General Exclusion Criteria:

* Participants with hematologic malignancies
* Concurrent administration of any other anti-cancer therapy (except male participants with prostate cancer receiving androgen blockade): Bisphosphonates and denosumab are allowed; Most recent anti-cancer therapy ≤28 days and have not recovered from the side effects, excluding alopecia; Radiation therapy within ≤14 days
* Active or untreated brain metastases
* History of carcinomatous meningitis
* Uncontrolled concurrent malignancy (early stage is allowed if not requiring active therapy or intervention)
* Pregnant or breastfeeding women, or intending to become pregnant during the study
* Any significant cardiovascular events within 6 months prior to study entry
* Pulmonary embolism within 30 days prior to study entry
* History or presence of clinically significant ventricular or atrial dysrhythmia >Grade 2 per NCI CTCAE v4.0
* Any other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or may interfere with the interpretation of study results
* Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol

Study-Drug Specific Exclusion Criteria:

Trastuzumab plus Pertuzumab

* Previous treatment with any HER2-targeted therapy

Erlotinib

* Non-small cell lung cancer (NSCLC) or pancreatic cancer identified by exon 19 deletions or exon 21 L858R substitution mutations
* EGFR amplifications in the absence of EGFR-activating mutations
* Cancers with exon 20 mutations
* Previous treatment with erlotinib or any other EGFR inhibitor
* Inability to swallow pills
* Refractory nausea and vomiting, malabsorption, external biliary shunt, or significant bowel resection that would preclude absorption of erlotinib

Vemurafenib plus Cobimetinib

* Malignant melanoma, papillary thyroid cancer, colorectal cancer, or hematologic malignancy including multiple myeloma
* LVEF below institutional lower level of normal (LLN) or below 50%, whichever is lower
* History of or evidence of retinal pathology on ophthalmologic examination that is considered a risk factor for neurosensory retinal detachment, retinal vein occlusion (RVO), or neovascular macular degeneration
* Presence of any of the following conditions, which are risk factors for RVO: Uncontrolled glaucoma with intraocular pressure >21 millimetres of mercury (mm Hg); Serum cholesterol ≥Grade 2; Hypertriglyceridemia ≥Grade 2; Hyperglycemia (fasting) ≥Grade 2; Grade ≥2 uncontrolled hypertension (participants with a history of hypertension controlled with anti-hypertensive medication to Grade </=1 are eligible)
* Prior or concurrent malignancy with known RAS mutation
* Previous treatment with vemurafenib or any other BRAF inhibitor (prior sorafenib is allowed)
* Previous treatment with cobimetinib or any other mitogen-activated protein/extracellular signal-regulated kinase (MEK) inhibitor
* Prior treatment with a RAF inhibitor
* Inability to swallow pills
* Refractory nausea and vomiting, malabsorption, external biliary shunt, or significant bowel resection that would preclude absorption of vemurafenib
* History of congenital long QT syndrome or mean (average of triplicate measurements) corrected QT (QTc) measured using Fridericia's method ≥450 millisecond (ms) at baseline or uncorrectable abnormalities in serum electrolytes (sodium, potassium, calcium, magnesium, phosphorus)

Vismodegib

* Basal cell carcinoma of the skin, medulloblastoma, small-cell lung cancer, or hematologic malignancies
* Previous treatment with vismodegib or any other hedgehog pathway inhibitor
* Inability to swallow pills
* Refractory nausea and vomiting, malabsorption, external biliary shunt, or significant bowel resection that would preclude absorption of vismodegib

Alectinib

* ALK-positive NSCLC, neuroblastoma, and childhood tumors
* Previous treatment with alectinib or any other ALK inhibitor
* Participants with symptomatic bradycardia
* Administration of strong/potent cytochrome P3A4 (CYP3A4) inhibitors or inducers within 14 days prior to the first dose of study treatment and while on treatment with alectinib
* Inability to swallow pills
* Refractory nausea and vomiting, malabsorption, external biliary shunt, or significant bowel resection that would preclude absorption of alectinib

Atezolizumab

* History of leptomeningeal disease
* Uncontrolled tumor pain
* Asymptomatic metastatic lesions that would likely cause functional deficits or intractable pain with further growth (e.g., epidural metastasis that is not currently associated with spinal cord compression) should be considered for loco-regional therapy if appropriate prior to enrollment
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently). Patients with indwelling catheters are allowed
* Uncontrolled or symptomatic hypercalcemia
* Previous treatment with atezolizumab or another programmed death-1 (PD-1)/PD-L1 inhibitor
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to biopharmaceutical agents produced in Chinese hamster ovary cells
* Known allergy or hypersensitivity to any component of the atezolizumab formulation
* Active or history of autoimmune disease or immune deficiency
* Prior allogeneic stem cell or solid organ transplantation
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan
* Positive human immunodeficiency virus (HIV) test, active hepatitis B virus (HBV) infection, active hepatitis C virus (HCV) infection or active tuberculosis
* Severe infection within 4 weeks prior to initiation of study treatment
* Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment
* Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction, or cerebrovascular accident within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina
* Major surgical procedure other than for diagnosis within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the course of the study
* Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during the course of the study or within 5 months after the final dose of atezolizumab
* History of other malignancy within 5 years prior to screening, with the exception of those with a negligible risk of metastasis or death, such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the participant at high risk from treatment complications
* Prior treatment with cluster of differentiation 137 (CD137) agonists or immune checkpoint blockade therapies
* Treatment with systemic immunostimulatory agents within 4 weeks or five half-lives of the drug (whichever is longer) prior to randomization
* Treatment with systemic immunosuppressive medication within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during the course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 673 (Actual)
Dates: Start 2014-04-14 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2023-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (60):
- United States (60):
  - Western Regional Medical Center at Cancer Treatment Centers of America, Goodyear, Arizona
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Highlands Oncology Group, Springdale, Arkansas
  - Science 37, Inc, Culver City, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Moores UCSD Cancer Center; Dept Clinical Trials Office, La Jolla, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Stanford Comprehensive Cancer Center, Stanford, California
  - Kaiser Permanente - Vallejo, Vallejo, California
  - University of Colorado, Aurora, Colorado
  - SCRI Florida Cancer Specialists South, Fort Myers, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Florida Hospital Cancer Inst; Memorial System Onc Clin Rsch, Orlando, Florida
  - Florida Cancer Specialist, North Region, St. Petersburg, Florida
  - Florida Cancer Specialists, Research Department, West Palm Beach, Florida
  - University Cancer & Blood Center, LLC; Research, Athens, Georgia
  - Northeast Georgia Medical Center; Oncology Research Dept-5C, Gainesville, Georgia
  - Southeastern Regional Medical Center, Inc., Newnan, Georgia
  - Northwestern University; Robert H. Lurie Comp Can Ctr; Northwestern Medicine Development Inst, Chicago, Illinois
  - University Of Chicago Medical Center; Section Of Hematology/Oncology, Chicago, Illinois
  - Midwestern Regional Med Center, Zion, Illinois
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Mayo Foundation, Rochester, Minnesota
  - Research Medical Center - Antibiotic Research Associates, Inc., Kansas City, Missouri
  - Memorial Sloan Kettering - Monmouth, Middletown, New Jersey
  - University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico
  - University of New Mexico Comprehensive Cancer Center - Albuquerque Cedar Street; Drug Shipment, Albuquerque, New Mexico
  - University of New Mexico Comprehensive Cancer Center - Albuquerque Lang NE; Drug Shipment, Albuquerque, New Mexico
  - University of New Mexico, Albuquerque, New Mexico
  - San Juan Oncology Associates, Farmington, New Mexico
  - Memorial Sloan Kettering Cancer Center at Westchester, Harrison, New York
  - Weill Cornell Univ Medical Ctr; Breast Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center; Herbert Irving Pavillion, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Univ No Carolina School of Med; Physicians Office Bldg, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest Univ Health Svcs; Internal Medicine, Winston-Salem, North Carolina
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Oncology Hematology Care Inc, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Providence Portland Medical Center, Portland, Oregon
  - Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Eastern Regional Medical Ctr, Philadelphia, Pennsylvania
  - UPMC - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Abington Mem Hosp-Abington; Rose. Can Ctr,Gyn Onc Ins, Willow Grove, Pennsylvania
  - Sanford Cancer Cnt Onco Clinic, Sioux Falls, South Dakota
  - Sarah Cannon Research Institute / Tennessee Oncology, Chattanooga, Tennessee
  - West Clinic, Germantown, Tennessee
  - Tennessee Cancer Specialists, Knoxville, Tennessee
  - Tennessee Oncology - Nashville, Nashville, Tennessee
  - Vanderbilt Ingram Cancer Clinic, Nashville, Tennessee
  - The Center for Cancer and Blood Disorders - Fort Worth, Fort Worth, Texas
  - MD Anderson, Houston, Texas
  - Virginia Cancer Institute, Richmond, Virginia
  - Northwest Medical Specialties, Tacoma, Washington
  - University of Wisconsin, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient-level data through the request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/).
  For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/innovation/process/clinical-trials/data-sharing/).

REFERENCES:
- [Derived] Sweeney CJ, Hainsworth JD, Bose R, Burris HA, Kurzrock R, Swanton C, Friedman CF, Spigel DR, Szado T, Schulze K, Price R, Malato J, Lo AA, Levy J, Wang Y, Yu W, Meric-Bernstam F. MyPathway Human Epidermal Growth Factor Receptor 2 Basket Study: Pertuzumab + Trastuzumab Treatment of a Tissue-Agnostic Cohort of Patients With Human Epidermal Growth Factor Receptor 2-Altered Advanced Solid Tumors. J Clin Oncol. 2024 Jan 20;42(3):258-265. doi: 10.1200/JCO.22.02636. Epub 2023 Oct 4. PMID 37793085
- [Derived] Narita Y, Yoshimoto T, Namai T, Asakawa T, Kawakami S, Gower-Page C, Reyes-Rivera I, Patel A, Nakamura Y. Pertuzumab Plus Trastuzumab for Treatment-Refractory HER2-Amplified Metastatic Colorectal Cancer: Comparison of the MyPathway Trial With a Real-World External Control Arm. JCO Clin Cancer Inform. 2022 May;6:e2200022. doi: 10.1200/CCI.22.00022. PMID 35649212
- [Derived] Friedman CF, Hainsworth JD, Kurzrock R, Spigel DR, Burris HA, Sweeney CJ, Meric-Bernstam F, Wang Y, Levy J, Grindheim J, Shames DS, Schulze K, Patel A, Swanton C. Atezolizumab Treatment of Tumors with High Tumor Mutational Burden from MyPathway, a Multicenter, Open-Label, Phase IIa Multiple Basket Study. Cancer Discov. 2022 Mar 1;12(3):654-669. doi: 10.1158/2159-8290.CD-21-0450. PMID 34876409
- [Derived] Javle M, Borad MJ, Azad NS, Kurzrock R, Abou-Alfa GK, George B, Hainsworth J, Meric-Bernstam F, Swanton C, Sweeney CJ, Friedman CF, Bose R, Spigel DR, Wang Y, Levy J, Schulze K, Cuchelkar V, Patel A, Burris H. Pertuzumab and trastuzumab for HER2-positive, metastatic biliary tract cancer (MyPathway): a multicentre, open-label, phase 2a, multiple basket study. Lancet Oncol. 2021 Sep;22(9):1290-1300. doi: 10.1016/S1470-2045(21)00336-3. Epub 2021 Jul 30. PMID 34339623
- [Derived] Meric-Bernstam F, Hurwitz H, Raghav KPS, McWilliams RR, Fakih M, VanderWalde A, Swanton C, Kurzrock R, Burris H, Sweeney C, Bose R, Spigel DR, Beattie MS, Blotner S, Stone A, Schulze K, Cuchelkar V, Hainsworth J. Pertuzumab plus trastuzumab for HER2-amplified metastatic colorectal cancer (MyPathway): an updated report from a multicentre, open-label, phase 2a, multiple basket study. Lancet Oncol. 2019 Apr;20(4):518-530. doi: 10.1016/S1470-2045(18)30904-5. Epub 2019 Mar 8. PMID 30857956
- [Derived] Hainsworth JD, Meric-Bernstam F, Swanton C, Hurwitz H, Spigel DR, Sweeney C, Burris H, Bose R, Yoo B, Stein A, Beattie M, Kurzrock R. Targeted Therapy for Advanced Solid Tumors on the Basis of Molecular Profiles: Results From MyPathway, an Open-Label, Phase IIa Multiple Basket Study. J Clin Oncol. 2018 Feb 20;36(6):536-542. doi: 10.1200/JCO.2017.75.3780. Epub 2018 Jan 10. PMID 29320312

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Trastuzumab Plus Pertuzumab | Atezolizumab | Vemurafenib | Vemurafenib Plus Cobimetinib | Vismodegib | Alectinib | Erlotinib
Started | 357 | 175 | 55 | 15 | 37 | 21 | 13
Completed | 28 | 24 | 3 | 0 | 3 | 0 | 0
Not Completed | 329 | 151 | 52 | 15 | 34 | 21 | 13
Not completed — Death | 280 | 118 | 46 | 13 | 31 | 16 | 12
Not completed — Withdrawal by Subject | 21 | 13 | 3 | 2 | 2 | 3 | 0
Not completed — Lost to Follow-up | 21 | 5 | 1 | 0 | 1 | 2 | 0
Not completed — Reason Not Specified | 6 | 5 | 2 | 0 | 0 | 0 | 1
Not completed — Study Ended by Sponsor | 1 | 9 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrew informed consent before receiving study drug | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are provided for the safety population, which includes all participants who received at least one dose of study treatment. One participant who enrolled in the atezolizumab arm withdrew from the study before receiving any treatment and was therefore excluded.
Groups:
- Total: Total of all reporting groups
Arm/Group | Trastuzumab Plus Pertuzumab | Atezolizumab | Vemurafenib | Vemurafenib Plus Cobimetinib | Vismodegib | Alectinib | Erlotinib | Total
Number analyzed (Participants) | 357 | 174 | 55 | 15 | 37 | 21 | 13 | 672
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 201 | 77 | 32 | 6 | 15 | 11 | 6 | 348
  >=65 years | 156 | 97 | 23 | 9 | 22 | 10 | 7 | 324
Age, Customized [Mean (Standard Deviation); unit: Years] | 61.0 (12.06) | 65.1 (12.33) | 61.3 (11.15) | 63.2 (8.69) | 63.5 (11.41) | 63.5 (12.17) | 64.5 (13.41) | 62.4 (12.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 179 | 98 | 29 | 7 | 16 | 12 | 5 | 346
  Male | 178 | 76 | 26 | 8 | 21 | 9 | 8 | 326
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 15 | 3 | 1 | 1 | 0 | 1 | 40
  Not Hispanic or Latino | 320 | 152 | 48 | 12 | 36 | 20 | 12 | 600
  Unknown or Not Reported | 18 | 7 | 4 | 2 | 0 | 1 | 0 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 3 | 0 | 0 | 0 | 0 | 1 | 7
  Asian | 21 | 11 | 1 | 0 | 3 | 0 | 1 | 37
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 28 | 20 | 7 | 1 | 2 | 2 | 0 | 60
  White | 288 | 131 | 46 | 13 | 31 | 18 | 10 | 537
  More than one race | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 16 | 8 | 1 | 1 | 1 | 1 | 1 | 29

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in All Tumor-Pathway Cohorts With Overall Response, as Assessed by the Investigator
Description: The Objective Response Rate (ORR) is defined as the percentage of patients whose best response on or before the first occurrence of disease progression is a complete response (CR) or partial response (PR). Tumor responses were assessed by investigators using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 for all arms.
Time Frame: From the date of first study treatment until disease progression or death from any cause, whichever occurs first (72.1 months)
Population: The efficacy evaluable population included all participants who received at least one dose of each drug for their assigned treatment regimen. The population includes the treated participants who have baseline tumor measurement and either have a post-baseline tumor measurement or have discontinued treatment for any reason.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Trastuzumab Plus Pertuzumab | Atezolizumab | Vemurafenib | Vemurafenib Plus Cobimetinib | Vismodegib | Alectinib | Erlotinib
Number analyzed (Participants) | 357 | 174 | 55 | 15 | 37 | 21 | 13
Percentage of Participants | 21.0 [16.9 to 25.6] | 19.5 [13.9 to 26.2] | 25.5 [14.7 to 39.0] | 33.3 [11.8 to 61.6] | 10.8 [3.0 to 25.4] | 14.3 [3.0 to 36.3] | 7.7 [0.2 to 36.0]

2. Primary Outcome: Percentage of Atezolizumab-Treated Participants With Tissue Tumor Mutational Burden (tTMB) ≥16 Mutations/Mb With Overall Response, as Assessed by the Independent Review Committee (IRC)
Description: The Objective Response Rate (ORR) is defined as the proportion of patients whose best response on or before the first occurrence of disease progression is a complete response (CR) or partial response (PR). Tumor responses were assessed by Independent Review Committee (IRC) using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Time Frame: From the date of first study treatment until disease progression or death from any cause, whichever occurs first (68.9 months)
Population: The efficacy evaluable population included all atezolizumab-treated participants with tumor mutation burden ≥16 Mutations/Mb and whose tumor responses were assessed by Independent Review Committee (IRC).
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Atezolizumab: Atezolizumab-treated participants with tissue TMB ( tTMB) ≥ 16 mutations/Mb (as assessed by FoundationOne or FoundationOne CDx). Participants received atezolizumab 1200 mg IV infusion every 3 weeks.
Arm/Group | Atezolizumab
Number analyzed (Participants) | 44
Percentage of Participants | 29.5 [16.8 to 45.2]

3. Secondary Outcome: Percentage of Participants With Disease Control
Description: Disease Control Rate (DCR) is defined as the proportion of patients whose best response is CR, PR or stable disease maintained more than 4 months (SD>4 months). Tumor responses were assessed by investigators using RECIST version 1.1 for all arms.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Trastuzumab Plus Pertuzumab | Atezolizumab | Vemurafenib | Vemurafenib Plus Cobimetinib | Vismodegib | Alectinib | Erlotinib
Number analyzed (Participants) | 357 | 174 | 55 | 15 | 37 | 21 | 13
Percentage of Participants | 41.5 [36.3 to 46.8] | 39.1 [31.8 to 46.8] | 34.5 [22.2 to 48.6] | 66.7 [38.4 to 88.2] | 16.2 [6.2 to 32.0] | 42.9 [21.8 to 66.0] | 23.1 [5.0 to 53.8]

4. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the time from the start of study treatment to the first occurrence of disease progression, or death, whichever occurs first. Tumor responses were assessed by investigators using RECIST version 1.1 for all arms.
Time Frame: From the date of first study treatment until disease progression as assessed by the investigator, or death from any cause, whichever occurs first (72.1 months)
Population: The efficacy evaluable population included all patients who received at least one dose of each drug for their assigned treatment regimen. The population includes the treated participants who have baseline tumor measurement and either have a post-baseline tumor measurement or have discontinued treatment for any reason.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trastuzumab Plus Pertuzumab | Atezolizumab | Vemurafenib | Vemurafenib Plus Cobimetinib | Vismodegib | Alectinib | Erlotinib
Number analyzed (Participants) | 357 | 174 | 55 | 15 | 37 | 21 | 13
Months | 2.8 [2.7 to 3.4] | 2.7 [1.6 to 3.0] | 3.1 [1.8 to 5.5] | 8.2 [3.9 to 19.5] | 1.8 [1.6 to 1.8] | 3.2 [1.7 to 6.6] | 1.8 [1.0 to 8.8]

5. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS, months) is defined as the time from the date of the first study treatment (Day 1) to the date of death from any cause.
Time Frame: 87.5 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trastuzumab Plus Pertuzumab | Atezolizumab | Vemurafenib | Vemurafenib Plus Cobimetinib | Vismodegib | Alectinib | Erlotinib
Number analyzed (Participants) | 357 | 174 | 55 | 15 | 37 | 21 | 13
Months | 10.1 [8.7 to 11.7] | 13.5 [11.2 to 17.4] | 10.6 [5.2 to 13.5] | 15.6 [6.8 to 27.9] | 9.8 [4.0 to 13.4] | 14.1 [8.7 to 25.6] | 7.7 [2.2 to 15.0]

6. Secondary Outcome: Duration of Response (DoR)
Description: Duration of Response (DoR) is defined as the time from the date of first documented response (CR or PR) to date of first occurrence of disease progression as determined by the investigator, or death from any cause, whichever occurs first.
Time Frame: From the date of first documented response (complete response [CR] or partial response [PR]) to the time of disease progression or death from any cause, whichever occurs first (70.8 months)
Population: Efficacy evaluable population who have achieved a complete or partial response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trastuzumab Plus Pertuzumab | Atezolizumab | Vemurafenib | Vemurafenib Plus Cobimetinib | Vismodegib | Alectinib | Erlotinib
Number analyzed (Participants) | 75 | 34 | 14 | 5 | 4 | 3 | 1
Months | 7.3 [5.8 to 9.3] | 32.1 [6.9 to NA] — The upper 95% confidence limit of median is not estimable due to insufficient number of events (disease progression/death) below 50th percentile of Kaplan-Meier curve | 6.0 [3.7 to 11.1] | 17.2 [7.4 to NA] — The upper 95% confidence limit of median is not estimable due to insufficient number of events (disease progression/death) below 50th percentile of Kaplan-Meier curve | 14.1 [6.5 to NA] — The upper 95% confidence limit of median is not estimable due to insufficient number of events (disease progression/death) below 50th percentile of Kaplan-Meier curve | 6.6 [6.0 to NA] — The upper 95% confidence limit of median is not estimable due to insufficient number of events (disease progression/death) below 50th percentile of Kaplan-Meier curve | 8.3 [NA to NA] — There was only one participant in this arm, therefore there are too few participants to calculate confidence intervals.

7. Secondary Outcome: Number of Participants With Adverse Events
Description: Incidence, nature, and severity of Adverse Events (AE), per the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03 (NCI CTCAE v4.03) for participants enrolled prior to Version 6 of the protocol. The NCI CTCAE (v5.0) grading scale was used for assessing AE severity for participants enrolled under Version 6 of the protocol and subsequent versions.
Time Frame: From first study treatment administration to 30 days (45 days for vismodegib, 90 days for atezolizumab) after the last dose (up to approximately 6.3 years)
Population: The safety (SAF) population is defined as enrolled patients who receive at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Trastuzumab Plus Pertuzumab | Atezolizumab | Vemurafenib | Vemurafenib Plus Cobimetinib | Vismodegib | Alectinib | Erlotinib
Number analyzed (Participants) | 357 | 174 | 55 | 15 | 37 | 21 | 13
Participants
  With at least one AE | 334 | 162 | 54 | 15 | 35 | 21 | 12
  With at least one SAE | 95 | 62 | 21 | 11 | 13 | 7 | 3
  With at least one Grade 3-5 AE | 146 | 97 | 37 | 12 | 21 | 11 | 4
  With at least one Related AE | 261 | 104 | 49 | 13 | 26 | 19 | 9
  With at least one Related SAE | 17 | 14 | 6 | 5 | 2 | 1 | 0
  With at least one Grade 3-5 related AE | 43 | 25 | 25 | 6 | 8 | 4 | 1
  With at least one non-serious AESI | 5 | 9 | 3 | 3 | 0 | 0 | 0
  With at least one AE leading to study drug withdrawn | 17 | 15 | 10 | 3 | 1 | 0 | 1
  With at least one AE leading to study drug interruption | 79 | 45 | 27 | 11 | 11 | 6 | 4
  With at least one AE leading to study drug reduction | 3 | 1 | 28 | 3 | 0 | 4 | 0
  With at least one AE leading to death | 13 | 5 | 2 | 2 | 1 | 0 | 1

ADVERSE EVENTS:
Time Frame: In the AE section, AE timeframe was from first study treatment administration to 30 days (45 days for vismodegib, 90 days for atezolizumab) after the last dose (up to approximately 6.3 years).
Description: The incidence, nature, and severity of Adverse Events (AE) and Serious Adverse Events (SAE) were reported, with severity determined according to NCI CTCAE v5.0 of the safety population, defined as all randomized participants who received ≥1 dose of study treatment.
Arm/Group | Trastuzumab Plus Pertuzumab | Atezolizumab | Vemurafenib | Vemurafenib Plus Cobimetinib | Vismodegib | Alectinib | Erlotinib
All-Cause Mortality (participants affected / at risk) | 285/357 | 118/174 | 46/55 | 13/15 | 31/37 | 16/21 | 12/13
Serious Adverse Events (participants affected / at risk) | 95/357 | 62/174 | 21/55 | 11/15 | 13/37 | 7/21 | 3/13
Other Adverse Events (participants affected / at risk) | 313/357 | 147/174 | 50/55 | 12/15 | 30/37 | 20/21 | 11/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab Plus Pertuzumab (N=357) | Atezolizumab (N=174) | Vemurafenib (N=55) | Vemurafenib Plus Cobimetinib (N=15) | Vismodegib (N=37) | Alectinib (N=21) | Erlotinib (N=13)
Anaemia (Blood and lymphatic system disorders) | 5 | 1 | 1 | 0 | 0 | 1 | 0
Anaemia of malignant disease (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Stress cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wolff-Parkinson-White syndrome (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 3 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 1 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Enterovesical fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 3 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 0 | 1 | 0
Obstruction gastric (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 6 | 3 | 0 | 3 | 2 | 0 | 1
Superior mesenteric artery syndrome (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 2 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Death (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 2 | 1 | 2 | 0 | 0 | 0
Sudden death (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Covid-19 pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Cholangitis infective (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium colitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Device related infection (Infections and infestations) | 3 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal viral (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Kidney infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Liver abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ophthalmic herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Perirectal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 4 | 5 | 2 | 0 | 2 | 0 | 1
Pneumonia aspiration (Infections and infestations) | 1 | 2 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 5 | 4 | 1 | 2 | 1 | 0 | 0
Sialoadenitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Soft tissue infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 5 | 2 | 2 | 1 | 0 | 0 | 0
Urinary tract infection bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection pseudomonal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Vascular device infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 5 | 0 | 0 | 0 | 0 | 0 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 1 | 0 | 0 | 2 | 0 | 0 | 0
International Normalised Ratio increased (Investigations) | 1 | 0 | 0 | 0 | 2 | 0 | 0
Liver function test increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 2 | 0 | 0 | 1 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Central nervous system lesion (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerebrospinal fluid leakage (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Dementia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Embolic cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Embolic stroke (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 3 | 2 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 4 | 4 | 1 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Autoimmune lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 2 | 1 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 1 | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Embolism (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab Plus Pertuzumab (N=357) | Atezolizumab (N=174) | Vemurafenib (N=55) | Vemurafenib Plus Cobimetinib (N=15) | Vismodegib (N=37) | Alectinib (N=21) | Erlotinib (N=13)
Anaemia (Blood and lymphatic system disorders) | 63 | 27 | 10 | 2 | 5 | 4 | 3
Abdominal distension (Gastrointestinal disorders) | 18 | 8 | 1 | 1 | 2 | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 43 | 25 | 6 | 5 | 1 | 4 | 1
Constipation (Gastrointestinal disorders) | 37 | 23 | 9 | 3 | 6 | 7 | 0
Diarrhoea (Gastrointestinal disorders) | 129 | 35 | 13 | 7 | 9 | 3 | 6
Nausea (Gastrointestinal disorders) | 80 | 40 | 21 | 8 | 8 | 6 | 4
Vomiting (Gastrointestinal disorders) | 47 | 26 | 13 | 6 | 2 | 1 | 1
Chills (General disorders) | 46 | 6 | 2 | 2 | 0 | 1 | 1
Fatigue (General disorders) | 105 | 46 | 29 | 7 | 14 | 7 | 5
Oedema peripheral (General disorders) | 26 | 14 | 5 | 6 | 6 | 7 | 0
Pyrexia (General disorders) | 36 | 16 | 4 | 5 | 2 | 1 | 4
Urinary tract infection (Infections and infestations) | 26 | 16 | 1 | 3 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 51 | 10 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 26 | 10 | 4 | 1 | 1 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 27 | 14 | 8 | 0 | 2 | 2 | 1
Blood alkaline phosphatase increased (Investigations) | 37 | 13 | 8 | 3 | 5 | 3 | 0
Blood bilirubin increased (Investigations) | 20 | 8 | 8 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 18 | 15 | 4 | 1 | 1 | 3 | 0
Weight decreased (Investigations) | 29 | 18 | 8 | 3 | 5 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 52 | 22 | 10 | 5 | 5 | 3 | 6
Dehydration (Metabolism and nutrition disorders) | 12 | 21 | 6 | 4 | 1 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 15 | 13 | 3 | 1 | 3 | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 29 | 4 | 5 | 2 | 3 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 21 | 24 | 4 | 0 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 44 | 22 | 18 | 4 | 2 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 32 | 22 | 7 | 1 | 2 | 6 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 23 | 1 | 0 | 1 | 7 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 16 | 16 | 6 | 2 | 5 | 4 | 2
Dizziness (Nervous system disorders) | 15 | 16 | 2 | 0 | 1 | 2 | 0
Headache (Nervous system disorders) | 27 | 21 | 8 | 0 | 3 | 2 | 1
Insomnia (Psychiatric disorders) | 27 | 6 | 4 | 1 | 2 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 44 | 29 | 6 | 2 | 1 | 3 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 41 | 20 | 6 | 2 | 4 | 5 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 25 | 5 | 7 | 2 | 2 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 35 | 20 | 4 | 2 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 38 | 5 | 11 | 4 | 2 | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 11 | 11 | 13 | 2 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-12-17): https://cdn.clinicaltrials.gov/large-docs/41/NCT02091141/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-17): https://cdn.clinicaltrials.gov/large-docs/41/NCT02091141/SAP_001.pdf